CLINICAL TRIAL: NCT01196182
Title: Congenital Heart Disease GEnetic NEtwork Study (CHD GENES)
Acronym: CHD GENES
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 701; 5U01HL098188-03 (NIH); U01HL098188 (NIH); U01HL098147 (NIH); U01HL098163 (NIH); U01HL098153 (NIH); U01HL098123 (NIH); U01HL098162 (NIH)
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Congenital Heart Defects
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood; possibly saliva and tissue.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Congenital heart defects (CHD) are the most common major human birth malformation, affecting ~8 per 1,000 live births. CHD are associated with significant morbidity and mortality, and are second only to infectious diseases in contributing to the infant mortality rate. Current understanding of the etiology of pediatric cardiovascular disorders is limited.

The Congenital Heart Disease GEnetic NEtwork Study (CHD GENES) is a multi-center, prospective observational cohort study. Participants will be recruited from the Pediatric Cardiac Genomics Consortium's (PCGC) centers of the NHLBI-sponsored Bench to Bassinet (B2B) Program. Biological specimens will be obtained for genetic analyses, and phenotype data will be collected by interview and from medical records. State-of-the-art genomic technologies will be used to identify common genetic causes of CHD and genetic modifiers of clinical outcome.

To accomplish this, the PCGC will develop and maintain a biorepository of specimens (DNA) and genetic data, along with detailed, phenotypic and clinical outcomes data in order to investigate relationships between genetic factors and phenotypic and clinical outcomes in congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

• Signed consent form

Exclusion Criteria:

* Isolated patent foramen ovale
* Isolated prematurity-associated patent ductus arteriosus

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: While all patients with pediatric cardiovascular disease and adults with congenital heart disease are of interest, the study will initially focus on four CHD anatomic classifications:
  * Atrial septal defects
  * Conotruncal abnormalities
  * Left-sided obstructive lesions
  * Heterotaxy
  Whenever possible, the study will recruit "trios" of participants--children, mothers and fathers-- as well as extended family members when appropriate and feasible.
Sampling Method: Non-Probability Sample
Enrollment: 32000 (Estimated)
Dates: Start 2010-11-15 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Roberts, MD, Principal Investigator — Childrens Hospital Boston; Christine Seidman, MD, Principal Investigator — Harvard Medical School, Boston MA; Bruce Gelb, MD, Principal Investigator — Mt Sinai School of Medicine, New York NY; Martina Brueckner, MD, Principal Investigator — Yale University; Martin Tristani-Firouzi, MD, Principal Investigator — University of Utah; Yufeng Shen, PhD, Principal Investigator — Columbia University Medical Center, New York NY; Shuo Wang, MD, Principal Investigator — Children's Los Angeles
Locations (15):
- United States (14):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Michigan Health, Ann Arbor, Michigan
  - Cohen Children's Medical Center New York, New Hyde Park, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Children's Hospital Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- University College London, London, United Kingdom

REFERENCES:
- [Derived] Jang MY, Patel PN, Pereira AC, Willcox JAL, Haghighi A, Tai AC, Ito K, Morton SU, Gorham JM, McKean DM, DePalma SR, Bernstein D, Brueckner M, Chung WK, Giardini A, Goldmuntz E, Kaltman JR, Kim R, Newburger JW, Shen Y, Srivastava D, Tristani-Firouzi M, Gelb BD, Porter GA Jr, Seidman CE, Seidman JG. Contribution of Previously Unrecognized RNA Splice-Altering Variants to Congenital Heart Disease. Circ Genom Precis Med. 2023 Jun;16(3):224-231. doi: 10.1161/CIRCGEN.122.003924. Epub 2023 May 11. PMID 37165897
- [Derived] Morton SU, Pereira AC, Quiat D, Richter F, Kitaygorodsky A, Hagen J, Bernstein D, Brueckner M, Goldmuntz E, Kim RW, Lifton RP, Porter GA Jr, Tristani-Firouzi M, Chung WK, Roberts A, Gelb BD, Shen Y, Newburger JW, Seidman JG, Seidman CE. Genome-Wide De Novo Variants in Congenital Heart Disease Are Not Associated With Maternal Diabetes or Obesity. Circ Genom Precis Med. 2022 Apr;15(2):e003500. doi: 10.1161/CIRCGEN.121.003500. Epub 2022 Feb 7. PMID 35130025
- [Derived] Oluwafemi OO, Musfee FI, Mitchell LE, Goldmuntz E, Xie HM, Hakonarson H, Morrow BE, Guo T, Taylor DM, McDonald-McGinn DM, Emanuel BS, Agopian AJ. Genome-Wide Association Studies of Conotruncal Heart Defects with Normally Related Great Vessels in the United States. Genes (Basel). 2021 Jul 1;12(7):1030. doi: 10.3390/genes12071030. PMID 34356046
- [Derived] Lahrouchi N, Postma AV, Salazar CM, De Laughter DM, Tjong F, Piherova L, Bowling FZ, Zimmerman D, Lodder EM, Ta-Shma A, Perles Z, Beekman L, Ilgun A, Gunst Q, Hababa M, Skoric-Milosavljevic D, Stranecky V, Tomek V, de Knijff P, de Leeuw R, Robinson JY, Burn SC, Mustafa H, Ambrose M, Moss T, Jacober J, Niyazov DM, Wolf B, Kim KH, Cherny S, Rousounides A, Aristidou-Kallika A, Tanteles G, Ange-Line B, Denomme-Pichon AS, Francannet C, Ortiz D, Haak MC, Ten Harkel AD, Manten GT, Dutman AC, Bouman K, Magliozzi M, Radio FC, Santen GW, Herkert JC, Brown HA, Elpeleg O, van den Hoff MJ, Mulder B, Airola MV, Kmoch S, Barnett JV, Clur SA, Frohman MA, Bezzina CR. Biallelic loss-of-function variants in PLD1 cause congenital right-sided cardiac valve defects and neonatal cardiomyopathy. J Clin Invest. 2021 Mar 1;131(5):e142148. doi: 10.1172/JCI142148. PMID 33645542
- [Derived] Sharma A, Wasson LK, Willcox JA, Morton SU, Gorham JM, DeLaughter DM, Neyazi M, Schmid M, Agarwal R, Jang MY, Toepfer CN, Ward T, Kim Y, Pereira AC, DePalma SR, Tai A, Kim S, Conner D, Bernstein D, Gelb BD, Chung WK, Goldmuntz E, Porter G, Tristani-Firouzi M, Srivastava D, Seidman JG, Seidman CE; Pediatric Cardiac Genomics Consortium. GATA6 mutations in hiPSCs inform mechanisms for maldevelopment of the heart, pancreas, and diaphragm. Elife. 2020 Oct 15;9:e53278. doi: 10.7554/eLife.53278. PMID 33054971
- [Derived] Boskovski MT, Homsy J, Nathan M, Sleeper LA, Morton S, Manheimer KB, Tai A, Gorham J, Lewis M, Swartz M, Alfieris GM, Bacha EA, Karimi M, Meyer D, Nguyen K, Bernstein D, Romano-Adesman A, Porter GA Jr, Goldmuntz E, Chung WK, Srivastava D, Kaltman JR, Tristani-Firouzi M, Lifton R, Roberts AE, Gaynor JW, Gelb BD, Kim R, Seidman JG, Brueckner M, Mayer JE Jr, Newburger JW, Seidman CE. De Novo Damaging Variants, Clinical Phenotypes, and Post-Operative Outcomes in Congenital Heart Disease. Circ Genom Precis Med. 2020 Aug;13(4):e002836. doi: 10.1161/CIRCGEN.119.002836. Epub 2020 Jun 30. PMID 32812804
- See also: Click here for more information about the entire Bench to Bassinet program. — http://www.benchtobassinet.org